CLINICAL TRIAL: NCT00190580
Title: Effects of Valsartan on the Progression of Renal and Cardiovascular Disease - Kanagawa Valsartan Trial (KVT)
Brief Title: Kanagawa Valsartan Trial (KVT): Effects of Valsartan on Renal and Cardiovascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KVT-Study Group (Other)
Collaborators: Tokai University (Other); Yokohama City University (Other); Showa University (Other); Kitasato University (Other); St. Marianna University School of Medicine (Other)
Responsible Party: Principal Investigator, Kenjiro Kimura, Professor of St. Marianna University School of Medicine, KVT-Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 620
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: CKD; chronic kidney disease; hypertension; angiotensin II receptor blocker; cardiovascular disease; valsartan; KVT
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Cardiovascular Diseases | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: valsartan; Drug: Conventional antihypertensive drugs
- 2 (Experimental)
  Interventions: Drug: Conventional antihypertensive drugs

INTERVENTIONS:
Drug: valsartan — valsartan, dosage from 20mg to 180mg, once or twice a day plus conventional antihypertensive drugs
  Other Names: Diovan 40mg or Diovan 80mg
  Arms: 1
Drug: Conventional antihypertensive drugs — Conventional antihypertensive drugs including calcium channel blockers, diuretics, angiotensin converting enzyme inhibitors and/or beta-blockers
  Other Names: any antihypertensive drug except ARB

SUMMARY:
The purpose of this study is to prove the hypothesis that the progression of renal and cardiovascular disease is more efficiently prevented when the angiotensin II receptor blocker valsartan is added to conventional antihypertensive therapy.

DETAILED DESCRIPTION:
It is widely recognized that suppression of the renin-angiotensin system ameliorates progression of chronic kidney disease (CKD) and that CKD is an important risk factor for development of cardiovascular disease. However, it has not been fully clarified if amelioration of CKD leads to the lower incidence of cardiovascular disease. The purpose of this study is to determine whether the angiotensin II receptor antagonist valsartan, in combination with conventional antihypertensive therapy, will ameliorate progression of both CKD and cardiovascular disease. The primary outcome is courses of renal and cardiac function. The secondary outcome is a composite of a doubling of serum creatinine concentration, end-stage renal disease, myocardial infarction, coronary revascularization, stroke, hospitalization for unstable angina, hospitalization for heart failure or death from cardiovascular causes.

ELIGIBILITY:
Inclusion Criteria:

* CKD with serum creatinine more than 2.0 mg/dl
* Blood pressure more than 130/85 mmHg
* 20 years old or above

Exclusion Criteria:

* End-stage renal disease with maintenance dialysis
* Polycystic kidney disease
* Collagen disease
* Malignant or accelerated hypertension

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2003-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Course of renal and cardiac function | every month for renal function and every year for cardiac function

SECONDARY OUTCOMES:
Doubling of serum creatinine concentration | every month
End-stage renal disease | anytime when it occurs.
Myocardial infarction | anytime when it occurs.
Coronary revascularization | anytime when it occurs.
Stroke | anytime when it occurs
Hospitalization for unstable angina | anytime when it occurs.
Hospitalization for heart failure | anytime when it occurs.
Death from cardiovascular causes | anytime when it occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Kenjiro Kimura, MD, PhD, Study Chair — St. Marianna University School of Medicine
Locations (1):
- St. Marianna University School of Medicine, Kawasaki, Kanagawa, Japan